CLINICAL TRIAL: NCT03374163
Title: Effect Of Intravenous IntralipidTherapyon Pregnancy Outcome in Women With History of Recurrent Implantation Failure Undergoing Intracytoplasmic Sperm Injection-Embryo Transfer Cycle: A Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, jawharah ali alzebidi, fellow, King Fahad Medical City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-442
Record Dates: First submitted 2017-12-05; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Infertility Due to Nonimplantation
Keywords: infertility , implantion failure, intracytoplasmic sperm injection
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: To evaluate the effect ofempiricintralipidinfusion therapy on pregnancy outcomes in patient withunexplained recurrentimplantation failure (RIF) undergoIntracytoplasmic sperm injection (ICSI).
  A total of 142 patients with history of unexplained RIF3 or more cycles were included in the study. Patient were randomized into two groups, study group (n=71) and control group (n=71). The study groupreceivedintralipid 20%infusionon the day of embryo transfer (ET) and a second dose on the day of pregnancy test. The control group underwent ET without intralipidinfusion.Allpatientswereclosely monitored for any side effectsincluding allergic reactions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- treatment group who recived intralipid (Experimental): 71 patients who recived intralipid on day of embryo transfer day, pregnancy day.
  Interventions: Drug: intralipid 20%
- control group (No Intervention): 71 patient not recived intralipid

INTERVENTIONS:
Drug: intralipid 20% — milky soulation for energey supplement.
  Arms: treatment group who recived intralipid

SUMMARY:
To evaluate the effect ofempiricintralipidinfusion therapy on pregnancy outcomes in patient withunexplained recurrentimplantation failure (RIF) undergoIntracytoplasmic sperm injection (ICSI).

DETAILED DESCRIPTION:
the aim to evaluate the effect ofempiricintralipidinfusion therapy on pregnancy outcomes in patient withunexplained recurrentimplantation failure (RIF) undergoIntracytoplasmic sperm injection (ICSI).

A total of 142 patients with history of unexplained RIF3 or more cycles were included in the study. Patient were randomized into two groups, study group (n=71) and control group (n=71). The study groupreceivedintralipid 20%infusionon the day of embryo transfer (ET) and a second dose on the day of pregnancy test. The control group underwent ET without intralipidinfusion.Allpatientswereclosely monitored for any side effectsincluding allergic reactions.

ELIGIBILITY:
Inclusion Criteria:

* age < 42 years
* BMI < 30 kg/m2
* history of 3 or more recurrent implantation failure undergoing Intracytoplasmic Sperm Injection (ICSI ) cycle.

exclusion criteria

* women with medical contraindications of intralipidinfusion.
* uterine fibroid.
* endometrial polyp.
* endometriosis,hydrosalpinx.
* intrauterine adhesion and uterine anomalies.
* Women with positive thrombophilia screen.
* diminished ovarian reserve.
* severe male factor infertility .
* chronic medical illnesses which may contribute in impaired chance of pregnancy .

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — biologicaly female
Enrollment: 142 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 14 day post embryo transfer day
  number of patient with positive b-hcg level 14 day post embryo transfer day.over the study population number in study period.

SECONDARY OUTCOMES:
miscarrage rate | miscarrage before 20 week gestation
  number of patient with miscarrage over study population number in study period
live birth rate | delivery after 28 week gestation
  number of patient with delivery after 28 week gestation over study population number in study period.

CONTACTS AND LOCATIONS:
Overall Officials: solaiman s alobaid, MD, Principal Investigator — King Fahad Medical City

IPD SHARING:
Plan to Share IPD: Yes